CLINICAL TRIAL: NCT05693909
Title: An Open-label, Dose-escalation, Dose-finding, and Proof-of-concept Trial of SP-420 in Subjects With Transfusion-dependent β-thalassemia or Low-risk Myelodysplastic Syndromes
Brief Title: A Trial Testing SP-420 in Subjects With Transfusion-dependent β-thalassemia or Low-risk Myelodysplastic Syndromes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: P-SP420-THAL-01
Record Dates: First submitted 2022-12-22; First posted 2023-01-23 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Beta Thalassemia Major Anemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — SP-420

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1a-1b (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420
- Cohort 2a-2b (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420
- Cohort 3a-3b (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420
- 1c-1d (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420
- 2c-2d (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420
- 3c-3d (Experimental): SP-420 for 48 weeks
  Interventions: Drug: SP-420

INTERVENTIONS:
Drug: SP-420 — Capsules for oral intake

SUMMARY:
The goal of this clinical trial is to learn about SP-420 ability to remove iron from organs in subjects with transfusion-dependent β-thalassemia or transfusion-dependent low-risk myelodysplastic syndrome.

The main questions it aims to answer are:

* How efficient is SP-420 in cleaning iron from the liver?
* How is the safety and tolerability of ascending doses of SP-420?

Participants will:

* Take medication three times weekly
* Attend up to 20 site visits
* Undergo MRI scans

ELIGIBILITY:
Thalassemia cohorts:

Inclusion criteria:

* Women and men aged 18 years or older
* Transfusion-dependent β-thalassemia including HbE/β-thalassemia requiring iron chelation therapy (β-thalassemia with mutation and/or multiplication of α-globin is allowed)
* On a stable dose of iron chelation for at least 4 weeks prior to screening
* Weight ≥ 35kg at screening
* Transfusion iron overload
* Treated and followed for at least the past 6 months in a specialized centre

Exclusion criteria:

* β-thalassemia with the structural Hb variants HbS and HbC
* Current MDS
* Current biliary disorder
* Historic or ongoing clinically significant kidney disease
* Unable to undergo trial assessments including MRI e.g. due to claustrophobia in MRI scanner
* Pregnant or nursing women
* Men who do not agree to practice effective barrier contraception during the entire period

Myelodysplastic Syndromes Cohorts:

Inclusion criteria:

* Women and men aged 18 years or older
* Very low, low, or intermediate risk Myelodysplastic Syndrome according to IPSS-R
* Weight ≥ 35kg at screening
* Transfusion iron overload
* Treated and followed for at least the past 6 months at medical facilities experienced with MDS

Exclusion criteria:

* Therapy-related MDS or MDS with a known bone marrow fibrosis
* Diagnosis of decompensated liver cirrhosis
* Clinically significant kidney disease, either historic or ongoing
* Uncontrolled ischemic heart disease or uncontrolled arrythmia
* Uncontrolled hypertension
* Uncontrolled dyslipidaemia
* Uncontrolled Diabetes
* Major surgery within 8 weeks prior to screening
* Pregnant or nursing women
* Men who do not agree to practice effective barrier contraception during the entire period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
To establish dose-response relationship of SP-420 for 24 weeks in the treatment of subjects with transfusion-dependent β-thalassemia | 24 weeks
To assess the safety and tolerability of ascending doses of SP-420 after 12 weeks treatment of subjects with transfusion-dependent low-risk myelodysplastic syndrome | 12 weeks

SECONDARY OUTCOMES:
To assess the efficacy of SP-420 in clearing iron from the liver after 24 weeks treatment of subjects with transfusion-dependent β-thalassemia | 24 weeks
  Change in liver iron concentration (LIC) measured by R2-magnetic resonance imaging (MRI) from baseline to week 24
To assess the efficacy of SP-420 in clearing iron from the liver after 12 and 48 weeks treatment of subjects with transfusion-dependent β-thalassemia | 12 and 48 weeks
  Change in LIC measured by R2-MRI from baseline to week 12 and week 48
To assess the efficacy of SP-420 on serum (s-) ferritin | up to 48 weeks
  Change in s-ferritin from baseline to weeks 1, 2, 3, 4, 6, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
To assess the safety and tolerability of ascending doses of SP-420 | 48 weeks
  Type and incidence of adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Pharmacosmos Clinical and non-clinical Department, Study Director — Pharmacosmos A/S
Locations (1):
- Pharmacosmos Investigational Site, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No